| Trial Name: | 105 |
|---|---|
| Trial Title: | The effect of food on the oral bioavailability of AEF0117 in healthy volunteers |
| Protocol No.: | AEF0117-105 |
| IND Number.: | 126501 |

| Reference to version and date of protocol on which report is based | |
|---|---|
| Protocol version: | 2 |
| Protocol date: | 01 December 2022 |

| Date: | 19 January 2023 |
|----------|-----------------|
| Version: | 1.0 |

Performed by:



Performed for:





Study : 105


Date: 19JAN2023

## Index

| 1. | Approv | als (signatures) | 11 |
|-----|--------------|---------------------------------------------|----|
| 2. | Distrib | ution List | 12 |
| 3. | Docum | ent Version History | 12 |
| 4. | Introduction | | |
| 4.1 | Ba | Background and rationale13 | |
| 4.2 | Ob | jectives | 14 |
| | 4.2.1 | Primary objective | 14 |
| | 4.2.2 | Secondary objectives | 14 |
| | 4.2.3 | Exploratory objective | 14 |
| 5. | Change | es to the protocol | 14 |
| 6. | Clinica | l trial methodology | 15 |
| 6.1 | Stu | dy design | 15 |
| 6.2 | Ra | ndomization | 15 |
| 6.3 | Sample size | | |
| 6.4 | Inte | erim analyses | 16 |
| 7. | Genera | l statistical considerations | 16 |
| 7.1 | Stu | dy population | 16 |
| 7.2 | Ge | neral issues | 16 |
| 7.3 | Pre | esentation/Format of results | 16 |
| 7.4 | Lev | vel of significance | 17 |
| 7.5 | На | ndling of dropouts and missing data | 17 |
| 8. | Statisti | cal analysis | 17 |
| 8.1 | De | finitions of variables | 17 |
| 8.2 | Ну | pothesis and statistical methods | 18 |
| | 8.2.1 | Univariate analysis. Descriptive statistics | 18 |
| | 8.2.2 | Bivariate analysis | 19 |
| 8.3 | De | mographic and baseline characteristics | 19 |



Study: 105 Version: 1.0

Date: 19JAN2023

| 8.4 | Prir | mary analysis | 19 |
|------|---------|------------------------------------------------------|-----|
| 8.5 | Sed | condary pharmacokinetic analysis | 20 |
| 8.6 | Saf | ety and tolerability analysis | 20 |
| 8.7 | Exp | oloratory objective | 22 |
| 8.8 | Сог | ncomitant medication | 22 |
| 9. | Referer | nces | 22 |
| 10. | | to be presented in the report | |
| 10.1 | | alysis sets | |
| 10.2 | Des | scriptive analysis - SAF | 27 |
| | 10.2.1 | Screening visit (Day -28 to -2) | 27 |
| | 10.2.2 | Baseline (Day -1) | 49 |
| | 10.2.3 | Follow-up | 66 |
| 10.3 | Prir | mary objective | 69 |
| | 10.3.1 | Pharmacokinetic endpoints | 69 |
| 10.4 | Sed | condary objectives | 71 |
| | 10.4.1 | Pharmacokinetic secondary endpoints | 71 |
| | 10.4.2 | Safety endpoints - Adverse Events | 72 |
| | 10.4.3 | Safety endpoints - Treatment Emergent Adverse Events | 78 |
| | 10.4.4 | Safety endpoints - Vital Signs | 85 |
| | 10.4.5 | Safety endpoints - Electrocardiogram | 88 |
| 10.5 | Saf | ety analysis | 97 |
| | 10.5.1 | Laboratory parameters – SAF | 97 |
| | 10.5.2 | Physical examination - SAF | 105 |
| | 10.5.3 | C-SSRS | 107 |
| 10.6 | Cor | ncomitant medication | 110 |
| 10.7 | List | ings | 111 |



Study: 105


Date: 19JAN2023

| Table index | |
|---|---|
| <b>Table 1.1.1</b> | Analysis sets - Subjects recruited24 |
| <b>Table 1.1.2</b> | Visits - SAF |
| <b>Table 1.1.3</b> | End of study - SAF |
| <b>Table 2.1.1</b> | Demographic - SAF |
| <b>Table 2.1.2</b> | Sex, Ethnicity and Status - SAF |
| <b>Table 2.1.3</b> | Contraception - SAF |
| <b>Table 2.1.4</b> | Medical history - SAF |
| <b>Table 2.1.5</b> | Ongoing medical history - SAF |
| <b>Table 2.1.6</b> | Physical examination (Screening) - SAF |
| <b>Table 2.1.7</b> | Vital signs (Screening) - SAF |
| <b>Table 2.1.8</b> | Electrocardiogram (Normal/Abnormal) (Screening) - SAF |
| <b>Table 2.1.9</b> | Electrocardiogram (Screening) - SAF |
| Table 2.1.10 | C-SSRS (Screening) - SAF |
| Table 0.4.44 | Laboratory evaluation (Screening) - SAF |
| Table 2.1.11 | Laboratory evaluation (Octeering) - SAI |
| Table 2.1.12 | Percentage of numeric values and non-numeric values (Screening) - |
| | Percentage of numeric values and non-numeric values (Screening) - |
| Table 2.1.12 | |
| Table 2.1.12<br>SAF 38 | Percentage of numeric values and non-numeric values (Screening) - |
| Table 2.1.12<br>SAF 38<br>Table 2.1.13 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |
| Table 2.1.12<br>SAF 38<br>Table 2.1.13<br>Table 2.1.14 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |
| Table 2.1.12<br>SAF 38<br>Table 2.1.13<br>Table 2.1.14<br>Table 2.1.15 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |
| Table 2.1.12<br>SAF 38<br>Table 2.1.13<br>Table 2.1.14<br>Table 2.1.15<br>Table 2.1.16 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |
| Table 2.1.12<br>SAF 38<br>Table 2.1.13<br>Table 2.1.14<br>Table 2.1.15<br>Table 2.1.16 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |
| Table 2.1.12<br>SAF 38<br>Table 2.1.13<br>Table 2.1.14<br>Table 2.1.15<br>Table 2.1.16<br>Table 2.2.1 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |
| Table 2.1.12<br>SAF 38<br>Table 2.1.13<br>Table 2.1.14<br>Table 2.1.15<br>Table 2.1.16<br>Table 2.2.1<br>Table 2.2.2 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |
| Table 2.1.12<br>SAF 38<br>Table 2.1.13<br>Table 2.1.14<br>Table 2.1.15<br>Table 2.1.16<br>Table 2.2.1<br>Table 2.2.2<br>Table 2.2.3 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |
| Table 2.1.12 SAF 38 Table 2.1.13 Table 2.1.14 Table 2.1.15 Table 2.1.16 Table 2.2.1 Table 2.2.2 Table 2.2.3 Table 2.2.4 Table 2.2.5 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |
| Table 2.1.12 SAF 38 Table 2.1.13 Table 2.1.14 Table 2.1.15 Table 2.1.16 Table 2.2.1 Table 2.2.2 Table 2.2.3 Table 2.2.4 Table 2.2.5 Table 2.2.5 | Percentage of numeric values and non-numeric values (Screening) - Chemistry (Screening) - SAF |




Date : 19JAN2023

| Table | 2.2.10 | Hematology (Baseline) - SAF | 59 |
|---|---|---|---|
| Table | 2.2.11 | Coagulation (Baseline) - SAF | 61 |
| Table | 2.2.12 | Urinary analysis (Baseline) - SAF | 62 |
| Table | 2.3.1 | CRU discharge (24 hours) - SAF | 66 |
| Table | 2.3.2 | Tests (days 3,4,5,7,9,11) - SAF | 67 |
| Table | 2.3.3 | Weight and BMI (312 h) - SAF | 68 |
| Table | 2.3.4 | Pregnancy test (312 hours) - SAF | 68 |
| Table | 3.1.1 | Descriptive analysis of pharmacokinetic endpoints - PK | 69 |
| Table | 3.1.2 | Regression analysis of pharmacokinetic endpoints - PK | 70 |
| Table | 4.1.1 | Descriptive analysis of pharmacokinetic secondary endpoints - PK | 71 |
| Table | 4.2.1 | General summary of adverse events – SAF | 72 |
| Table | 4.2.2 | AE I (Fed) - SAF | 74 |
| Table | 4.2.3 | AE II (Fed) - SAF | 75 |
| Table | 4.2.4 | AE III (Fed) - SAF | 76 |
| Table | 4.2.5 | AE I (Fasting) - SAF | 77 |
| Table | 4.2.6 | AE II (Fasting) – SAF | 77 |
| Table | 4.2.7 | AE III (Fasting) - SAF | 77 |
| Table | 4.3.1 | General summary of treatment emergent adverse events – SAF | 78 |
| Table | 4.3.2 | TEAE I (Fed) - SAF | 80 |
| Table | 4.3.3 | TEAE II (Fed) - SAF | 81 |
| Table | 4.3.4 | TEAE III (Fed) - SAF | 82 |
| Table | 4.3.5 | TEAE III (Fed) - SAF | 83 |
| Table | 4.3.6 | TEAE I (Fasting) - SAF | 84 |
| Table | 4.3.7 | TEAE II (Fasting) – SAF | 84 |
| Table | 4.3.8 | TEAE III (Fasting) - SAF | 84 |
| Table | 4.4.1 | Time between evaluation and dose (hours) - SAF | 85 |
| Table | 4.4.2 | SBP - Supine (mmHg) - SAF | 87 |
| Table | 4.4.3 | DBP - Supine (mmHg) - SAF | 87 |
| Table | 4.4.4 | Heart rate - Supine (bpm) - SAF | 87 |
| Table | 4.4.5 | Oral temperature (°C) - SAF | 87 |
| Table | 4.5.1 | Electrocardiogram (Normal/Abnormal) - SAF | 88 |




Date: 19JAN2023

| Table | 4.5.2 | Time between ECG and dose (hours) - SAF | . 95 |
|-------|--------|-----------------------------------------------|------|
| Table | 4.5.3 | Heart rate (BPM) - SAF | . 96 |
| Table | 4.5.4 | PR intervals (ms) - SAF | . 96 |
| Table | 4.5.5 | QRS duration (ms) - SAF | . 96 |
| Table | 4.5.6 | QT interval (ms) - SAF | . 96 |
| Table | 4.5.7 | QTcF interval (ms) - SAF | . 96 |
| Table | 5.1.1 | Time between evaluation and dose (days) - SAF | . 97 |
| Table | 5.1.2 | Non numeric values – SAF | . 98 |
| Table | 5.1.3 | Chemistry - Albumin (g/dl) - SAF | . 99 |
| Table | 5.1.4 | Chemistry – ALP (U/L) - SAF | . 99 |
| Table | 5.1.5 | Chemistry - ALT (GPT) (U/L) - SAF | . 99 |
| Table | 5.1.6 | Chemistry - AST (GOT) (U/L) - SAF | . 99 |
| Table | 5.1.7 | Chemistry – Bicarbonate (mEq/L) - SAF | . 99 |
| Table | 5.1.8 | Chemistry – Blood urea nitrogen (mg/dL) - SAF | . 99 |
| Table | 5.1.9 | Chemistry - Calcium (mg/dL) - SAF | . 99 |
| Table | 5.1.10 | Chemistry - Total Cholesterol (mg/dL) - SAF | . 99 |
| Table | 5.1.11 | Chemistry - Creatinine (mg/dL) - SAF | . 99 |
| Table | 5.1.12 | Chemistry - CPK (U/L) - SAF | . 99 |
| Table | 5.1.13 | Chemistry - Glucose (mg/dL) - SAF | . 99 |
| Table | 5.1.14 | Chemistry - HDL (mg/dL) - SAF | . 99 |
| Table | 5.1.15 | Chemistry - LDL (mg/dL) - SAF | . 99 |
| Table | 5.1.16 | Chemistry - Phosphorus (mg/dL) - SAF | 100 |
| Table | 5.1.17 | Chemistry - Potassium (mmol/L) - SAF | 100 |
| Table | 5.1.18 | Chemistry – Total Bilirubin (mg/dL) - SAF | 100 |
| Table | 5.1.19 | Chemistry - Sodium (mmol/L) – SAF | 100 |
| Table | 5.1.20 | Chemistry – Total Protein (g/dL) – SAF | 100 |
| Table | 5.1.21 | Chemistry - Triglycerides (mg/dL) - SAF | 100 |
| Table | 5.1.22 | Chemistry – Uric acid (mg/dL) - SAF | 100 |
| Table | 5.1.23 | Hematology - Hematocrit (%)- SAF | 100 |
| Table | 5.1.24 | Hematology - Hemoglobin (g/dL) - SAF | 100 |
| Table | 5.1.25 | Hematology - MCV (fL) - SAF | 100 |




Date : 19JAN2023

| Table | 5.1.26 | Hematology - MCHC (g/L) - SAF | . 100 |
|-------|--------|----------------------------------------------|-------|
| Table | 5.1.27 | Hematology - Platelet count (x10^3 μL) - SAF | . 100 |
| Table | 5.1.28 | Hematology - RBC (x10^6 μL) - SAF | . 100 |
| Table | 5.1.29 | Hematology - WBC (x10^3 μL) - SAF | . 100 |
| Table | 5.1.30 | Hematology - Basophils (x10^3 μL) - SAF | . 100 |
| Table | 5.1.31 | Hematology - Eosinophils (x10^3 μL) - SAF | . 100 |
| Table | 5.1.32 | Hematology - Lymphocytes (x10^3 μL) - SAF | . 100 |
| Table | 5.1.33 | Hematology - Monocytes (x10^3 μL) - SAF | . 100 |
| Table | 5.1.34 | Hematology - Neutrophils (x10^3 μL) - SAF | . 100 |
| Table | 5.1.35 | Coagulation - INR - SAF | . 100 |
| Table | 5.1.36 | Coagulation - Prothrombine time (s) - SAF | . 100 |
| Table | 5.1.37 | Coagulation - aPTT (s) - SAF | . 100 |
| Table | 5.1.38 | Urine analysis – Color and appearance – SAF | . 101 |
| Table | 5.1.39 | Urine Analysis – ph - SAF | . 102 |
| Table | 5.1.40 | Urine analysis – Specific gravity – SAF | . 102 |
| Table | 5.1.41 | Urine Analysis - Glucose - SAF | . 103 |
| Table | 5.1.42 | Urine Analysis – Protein – SAF | . 104 |
| Table | 5.1.43 | Urine Analysis –Red blood cells – SAF | . 104 |
| Table | 5.1.44 | Urine Analysis – Leukocytes – SAF | . 104 |
| Table | 5.1.45 | Urine Analysis – Ketones – SAF | . 104 |
| Table | 5.1.46 | Urine Analysis –Bilirubin – SAF | . 104 |
| Table | 5.1.47 | Urine Analysis – Urobilinogen – SAF | . 104 |
| Table | 5.1.48 | Urine Analysis – Nitrite - SAF | . 104 |
| Table | 5.2.1 | Physical examination - SAF | . 105 |
| Table | 5.3.1 | C-SSRS - SAF | . 107 |
| Table | 6.1.1 | Previous concomitant medication | . 110 |
| Table | 612 | Concomitant medication during study | 110 |



Study : 105


Date: 19JAN2023

# Listing index

| Listing 7.1.1 | Discontinued subjects | 111 |
|---|---|---|
| Listing 7.1.2 | Protocol deviations | 111 |
| Listing 7.1.3 | Subjects excluded from population analysis | 111 |
| Listing 7.1.4 | Baseline data | 112 |
| Listing 7.1.5 | Prior concomitant medication | 112 |
| Listing 7.1.6 | Concomitant medication during study | 112 |
| Listing 7.1.7 | Adverse Events | 113 |
| Listing 7.1.8 | Serious adverse events | 113 |
| Listing 7.1.9 | Abnormal findings on physical examination | 114 |
| Listing 7.1.10 | Abnormal findings on vital signs, ECG and laboratory results | 114 |
| Listing 7.1.11 | COVID-19 tests | 114 |




Date: 19JAN2023

## **ABBREVATIONS AND DEFINITIONS**

| ABBREVAII | ONS AND DEFINITIONS |
|------------------|-----------------------------------------------------------|
| ACT | Anatomical Therapeutic Chemical |
| AE | Adverse Event |
| ALP | Alkaline Phosphatase |
| ALT (GPT) | Alanine transaminase |
| aPTT | Activated Partial Thromboplatin time |
| AST (GOT) | Aspartate Transaminase |
| AUC | Area Under the Curve |
| ВМІ | Body Mass Index |
| C <sub>24h</sub> | Observed plasma concentration 24 hours after dose |
| CB1 | Cannabinoid receptor type 1 |
| CI | Confidence Interval |
| CL/F | Apparent clearance |
| C <sub>max</sub> | Maximum observed plasma concentration |
| СРК | Creatine Phosphokinase |
| CRU | IMIM-Clinical Research Unit |
| CS | Clinically Significant |
| C-SSRS | Columbia Suicide Severity Rating Score |
| CUD | Cannabis User Disorder |
| CV | Coefficient of variation |
| DBP | Diastolic Blood Pressure |
| ECG | Electrocardiogram |
| FDA | Food and Drug Administration |
| FSH | Follicle-stimulating hormone |
| HDL | High-density Lipoprotein |
| IB | Investigator's Brochure |
| INR | International Normalized Ratio |
| INSERM | Institut National de la Santé et de la Recherche Médicale |
| LDL | Low-density Lipoprotein |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCV | Mean Corpuscular Volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCS | Non-clinically significant |
| PK | Pharmacokinetic(s) |
| PT | Preferred Term |
| Q1, Q3 | Quartiles 1 and 3 |
| QTcF | QT interval corrected |
| | • |



| Study : 105 |
|------------------|
| Date : 19IAN2023 |

| RBC | Red blood cell count |
|---|---|
| SAF | Safety analysis set |
| SAS® | Statistical Analysis System |
| SBP | Systolic Blood Pressure |
| sCB1-SSi | Synthetic signaling specific inhibitor of the CB1 receptor |
| SD | Standard Deviation |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TEAE | Treatment Emergent Adverse Event |
| THC | Tetrahydrocannabinol |
| t <sub>lag</sub> | Time to first quantifiable plasma concentration |
| T <sub>max</sub> | Time to observed maximum plasma concentration |
| Vd/F | Apparent volume of distribution |
| WBC | White blood cells |
| WHOdrug | World Health Organization-drug |



| Study : 105 |
|--------------|

Date: 19JAN2023

# 1. Approvals (signatures)

The signatures on this page indicate review and approval of the statistical analysis plan and referenced Sections.

| <u>Bioclever</u> | |
|---------------------------------------|-------|
| Written by: Josep Puig, Biostatiscian | |
| (Sig.) | Date: |
| Aelis Farma | |
| Approved by: Lasse Steen Ravn, MD | |
| (Sig.) | Date: |



| Study : 105 |
|------------------|
| Date : 19JAN2023 |

# 2. Distribution List

| Name | Function / Role | Office/Sponsor |
|----------------------|-----------------|----------------|
| Ghislaine Campistron | Sponsor | AELIS FARMA |
| Audrey Serpault | Sponsor | AELIS FARMA |
| Lasse Steen Ravn | Sponsor | AELIS FARMA |
| Arnau Lucas | CRO | Bioclever |

# 3. Document Version History

| Version | Effective Date | Significant Changes |
|---|---|---|
| 0.1 | 25 October 2022 | Minor changes. |
| 0.2 | 09 November 2022 | Minor changes. |
| 0.3 | 05 December 2022 | Minor changes. |
| 0.4 | 09 January 2023 | New protocol version. Urine collection for exploratory objective has been deleted. |
| 0.5 | 13 January 2023 | No changes. |




Date: 19JAN2023

# 4. Introduction

# 4.1 Background and rationale

Cannabis is the most widely used illicit drug with approximately 28 million individuals reporting past-month use [1], and 14% of those receiving substance use disorder treatment in the US reporting cannabis as their primary drug of abuse [2]. While psychotherapeutic approaches have some utility for treating Cannabis Use Disorder (CUD) [3, 4, 5, 6], the vast majority of patients have difficulty significantly reducing their use or achieving abstinence. Safe and effective medications to treat CUD are urgently needed [7, 8]. The overall goal of this clinical trial is to contribute to advancing a safe and effective pharmacotherapy for CUD along the FDA approval pipeline.

When the CB1 receptors are over-activated by very high doses of THC, quite higher than the doses of THC used by cannabis abusers, the concentration of the steroid hormone pregnenolone increases in the brain. Pregnenolone then binds to a specific site on the CB1 receptors, distinct for the one of CB1 agonists and THC, and acts as an endogenous signaling specific inhibitor of the CB1 receptors. However, pregnenolone does not modify the binding of CB1 agonists to the CB1 receptor. Despite this restricted molecular action, when pregnenolone is administered prior to the exposure to THC, it inhibits most of the THC-mediated behavioral effects in rodents and THC self-administration in non-human primates. Pregnenolone cannot be used as a pharmacological treatment because it is poorly bioavailable, has a very short half-life and is converted downstream to active steroids. Aelis Farma, in collaboration with researchers from the Institut National de la Santé et de la Recherche Médicale (INSERM), has developed a new pharmacological class, the synthetic signaling specific inhibitor of the CB1 receptor (sCB1-SSi), by modifying pregnenolone's chemical structure to prevent conversion to active steroids, and to increase absorption and biological stability while maintaining THC antagonism.

To date, 3 clinical studies have been completed with AEF0117 including 2 phase 1 studies in healthy volunteers (AEF0117-101 single ascending dose study and AEF0117-102, multiple ascending dose study), and a phase 2a trial in cannabis users (AEF0117-201). The phase 1 studies showed good safety and tolerability of AEF0117 in the dose range tested (0.2 mg as single dose and 0.6–6 mg/day as single and multiple doses) and the phase 2a trial found that the 1 mg/day dose of AEF0117 significantly reduced both the abuse-related subjective effects of cannabis and its self-administration, while the 0.06 mg dose did not. Importantly, AEF0117 was well tolerated in daily cannabis smokers, with no evidence of precipitated withdrawal, physical, or psychological discomfort. There were no SAEs and a limited number of TEAEs. These results confirm preclinical data showing that AEF0117 does not function as an orthosteric antagonist and does not produce any of the adverse effects associated with rimonabant. Thus, AEF0117 is to our knowledge the first medication to safely and robustly



| Study : 105 |
|--------------|

Date: 19JAN2023

attenuate the positive subjective and reinforcing effects of cannabis in participants with CUD. Further details are provided in the current edition of the IB [9].

In the 3 early studies conducted with AEF0117, AEF0117 was administered orally after a light breakfast. AEF0117 showed a good bioavailability and favorable, dose-proportional PK [9]. In this protocol, the effects of food on AEF0117 bioavailability in healthy volunteers will be investigated by comparing the rate and extent of AEF0117 absorption when 1 mg AEF0117 is administered in fed state versus fasting state.

The safety and tolerability of AE0117 has been demonstrated in the clinical studies conducted to date. This trial will provide data on the effect of food on the oral bioavailability of AEF0117 to support the next stage of the clinical development of the drug.

# 4.2 Objectives

## 4.2.1 Primary objective

To determine the bioavailability of orally administered AEF0117 after fed conditions relative to fasting conditions in healthy volunteers.

# 4.2.2 Secondary objectives

- To evaluate other PK parameters of AEF0117 in healthy volunteers.
- To evaluate safety and tolerability of a single dose of 1 mg AEF0117 in healthy volunteers.

# 4.2.3 Exploratory objective

To characterize potential metabolites regarding plasma PK.

# 5. Changes to the protocol

The protocol states "An analysis of variance model will be applied, with sequence, period, and state (fed, fasting) as factors". This is not a cross-over study for that reason period and sequence variables do not apply. The analysis of variance model has been changed for a t-test analysis (See section 8.4).



| Study : 105 |
|--------------|

Date: 19JAN2023

# 6. Clinical trial methodology

# 6.1 Study design

This is a single center, randomized, parallel-group, 2-arm, open-label, single-dose trial in healthy male and female volunteers aged 18–55 years, both inclusive.

The total trial duration for an individual participant will be up to 6 weeks (42 days) from screening (up to 28 days prior to dosing) to the final follow-up visit (14 days after dosing).

After screening, the trial includes 2 days where the participants are confined at the research facility, and thereafter 7 visits to the site (6 visits and a follow-up visit). Participants will stay in the research facility from the afternoon prior to dosing on Day 1 and until collection of the blood sample 24 hours after dosing (i.e., Day 2) and then be discharged. Participants will be asked to return to the research facility for collection of blood samples each morning on Days 3, 4, 5, 7, 9, and 11, and at the follow-up visit on Day 14.

On Day 1, eligible participants will be randomized and receive a single dose of 1 mg AEF0117 in fed or fasting condition, and serial blood samples will be collected up to 312 hours after dose administration

### 6.2 Randomization

All participants will be assigned a unique trial participant number at the trial-specific screening.

A computer-generated randomization schedule will be prepared by a statistician. Eligible participants will be randomly assigned to 1 of the 2 groups. Randomization will be with a block size of 2 and stratified by sex.

The 2 groups will be divided into smaller cohorts of at least 2 participants for operational reasons (adjusted to in clinic facilities) and each cohort will include a similar number of participants from each group (fed or fasting).



| Study : 105 |
|--------------|

Date: 19JAN2023

# 6.3 Sample size

The sample size has been chosen based on previous experience in phase 1 studies with AEF0117 where the CV was in the order of 0.3 for Cmax and AUC after single doses. It is anticipated that food slightly increases the absorption of AEF0117 and a true ratio of 1.25 is assumed. To allow for potential participants who dropout early, i.e., not allowing for estimation of Cmax and/or AUC0-t, 32 participants should be included. The power for showing that the upper bound of the 2-sided 90% CI of the geometric mean ratio is ≤1.75 is 90% with 14 participants per treatment group and 86% with 12 participants per group.

# 6.4 Interim analyses

Not applicable.

# 7. General statistical considerations

# 7.1 Study population

- <u>Safety analysis set (SAF)</u>: This set will include all randomized subjects in the study who recieved the study drug (AEF0117).
- Pharmacokinetic(s) analysis set (PK analysis set): This set will include all randomized subjects in the study who recieved the study drug (AEF0117) with sufficient and valid plasma drug concentration data to allow the determination of PK parameters (at least the 24-hour PK profile), without vomits within 3 hours after dose and without protocol deviations with significant influence on estimation of one or more PK parameter.

### 7.2 General issues

All data processing, summarization and analyses will be performed using SAS® version 9.4 or posterior.

### 7.3 Presentation/Format of results

Mean, median and standard deviation will be printed out to one more decimal place than the recorded data and rounded appropriately. Minimum and maximum values will be presented using the same number of decimal places as the recorded data. The number of subjects will be presented as a whole number.

Percentage values will be presented with one digit to the right of decimal point.

P-values will be presented to 4 decimal places (or as <0.0001 where appropriate).




Date: 19JAN2023

# 7.4 Level of significance

Statistical comparisons will be made using two sided tests at the  $\alpha$ =0.05 significance level unless specifically stated otherwise.

# 7.5 Handling of dropouts and missing data

No imputation method will be used.

# 8. Statistical analysis

### 8.1 Definitions of variables

- Age (years):

(Date of informed consent - Date of birth) / 365.25

- Duration of adverse events:

Duration (minutes) = (End time[hh:mm] and date - initial time[hh:mm] and date)

- Time between two events (hours, days and months):

Hours: (Most recent Date - Other Date) / 60 [Format date: Day/Month/Year, Hour:Minute]

Days: Most recent Date – Other Date [Format date: Day/Month/Year]

Months: (Most recent Date – Other Date) / 30.4375 [Format date: Day/Month/Year]

# C-SSRS:

### Categories:

Category 1 – Wish to be Dead

Category 2 – Non-specific Active Suicidal Thoughts

Category 3 – Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act

Category 4 - Active Suicidal Ideation with Some Intent to Act, without Specific Plan

Category 5 - Active Suicidal Ideation with Specific Plan and Intent

Category 6 - Preparatory Acts or Behavior

Category 7 - Aborted Attempt

Category 8 – Interrupted Attempt

Category 9 – Actual Attempt (non-fatal)

Category 10 - Completed Suicide (not included at screening and baseline visit)

Suicidal Ideation or Behavior:



| Study : 105 |
|------------------|
| Date : 19JAN2023 |

Yes: If any category = "Yes".

No: All categories = "No".

### Suicidal Ideation:

- Yes: If any category 1-5 = "Yes".

- No: All categories 1-5 = "No".

### Suicidal Behavior:

- Yes: If any category 6-10 = "Yes".

No: All categories 6-10 = "No".

All suicidal endpoints will be calculated before study (screening visit and baseline visit) and during study (study visits)

- Treatment Emergent Adverse Event (TEAE):

Adverse Events with an onset equal or posterior to IMP administration

- ECG parameters:

For each timepoint 3 ECGs will be performed. The results of them will be summarized as:

- o Normal/Abnormal:
  - Three Normal ECG -> "All normal"
  - One, two or three Abnormal ECG -> "Any Abnormal"
- Does the result meet the definition of adverse event? (Yes/No) [Overall ECG variable and per parameter variable (Heart rate, PR Inteval, QRS duration, QT interval, QTcF intervals)]:
  - Three "No" -> "All No"
  - One, two or three "Yes" -> "Any Yes"
- o Heart rate: Mean value of 3 ECGs.
- o PR interval: Mean value of 3 ECGs.
- o QRS duration: Mean value of 3 ECGs.
- o QT interval: Mean value of 3 ECGs.
- o QTcF intervals: Mean value of 3 ECGs.

# 8.2 Hypothesis and statistical methods

## 8.2.1 Univariate analysis. Descriptive statistics

Unless otherwise noted, all variables will be described according to their character as follows:



| | Study : 105 |
|---|--------------|
| _ | |

Date: 19JAN2023

- Categorical variables will be summarized using frequencies and percentages.
- Continuous variables will be summarized using measures of central tendency and dispersion: mean, standard deviation, median, 25% and 75% percentiles (Q1 and Q3) and extreme values (minimum and maximum).

## 8.2.2 Bivariate analysis

When it is of interest to answer the study objectives, the relationship between variables will be evaluated:

- For two categorical variables, contingency tables with the frequency in each category and the percentage by columns will be presented.
- For a numerical variable with a categorical, descriptive statistics will be presented by groups.

# 8.3 Demographic and baseline characteristics

Demographic data and baseline characteristics will be described following the methods that appear in section 8.2.

# 8.4 Primary analysis

Plasma PK parameters:

- Area under the concentration-time curve (AUC<sub>0-t</sub>, AUC<sub>0- $\infty$ </sub>) where t is the last or the latest timepoint observed.
- Observed maximum plasma concentration: C<sub>max</sub>.
- Time to observed maximum plasma concentration:  $T_{\text{max}}$ .
- Time lag (Time to first quantifiable plasma concentration): t<sub>lag</sub>.

PK analysis will consist of a non-compartmental evaluation of AEF0117 plasma concentration-time profiles to determine PK parameters using a validated program. PK analysis will be performed at PK lab before transferred for statistical analysis.

### For each PK parameter:

- A descriptive analysis by fed and fasting will be presented.
- A t-test will be fitted by using PROC TTEST (SAS) for all parameters except  $T_{\text{max}}$  and  $t_{\text{lag}}$ :
  - The natural logarithm transformation of each parameter will be the response variable.



| Study : | 105 |
|--------------|-------|
| Version | : 1.0 |
| Date : 19JAN | 2023 |

o Exploratory variable will be:

State: Fed / Fasting.

- A table with the t-test p-value, the exponential of estimated mean difference (Geometric mean ratio) and its 90% confidence interval will be presented.
- Relative bioavailability is the ratio of AUCs. The relative bioavailability of AEF0117 under fed conditions compared to under fasting condition will be assessed as negligeable during therapeutic use if the two-sided 90% CI of fed vs fasting is <= 1.75. Bioequivalence will be declared if the 90% CI is included in 0.8-1.25 range.

# 8.5 Secondary pharmacokinetic analysis

Plasma PK parameters:

- %AUCextrap
- Observed concentration 24 hours after dose: C<sub>24h</sub>.
- Terminal elimination half-life: t<sub>1/2</sub>.
- Apparent clearance: CL/F.
- Apparent volume of distribution: Vd/F.

A descriptive analysis by fed and fasting will be presented.

# 8.6 Safety and tolerability analysis

Safety and tolerability endpoints:

- Any AE per subject and state.
- Any TEAE per subject and state.
- Vital signs.
- ECG.
- Laboratory parameters (Hematology, Chemistry, Coagulation profile and urinanalysis).
- Physical examination
- C-SSRS.

A descriptive analysis by fed/fasting will be presented.

Frequency and percentage of subjects and number of AE and TEAE will be included, by the following variables:

- Severity: Mild, Moderate, Severe.
- Causality: Not related, Related.



| Study : 105 |
|--------------|

Date: 19JAN2023

- Action taken with study treatment: Dose not changed, drug withdrawn, drug interrupted, dose increased, dose reduced, not applicable, unknown.
- Outcome: Recovered/Resolved, Recovering/Resolving, Not recovered/Not resolved, Recovered/Resolved with sequelae, Fatal, Unknown
- Serious: Yes, No.
- Serious criteria: Death, Hospitalization or prolongation of existing hospitalization, Congenital anomaly or birth defect, Other medically important event, Life threatening, Significant disability/incapacity.

Also a descriptive analysis of AE and TEAE by System Organ Class and Preferred Term (codificated by the dictionary MedDRA version 25.0) will be presented.




Date: 19JAN2023

# 8.7 Exploratory objective

The exploratory analysis will be performed in the future. The analysis will be included in another document.

### 8.8 Concomitant medication

The concomitant medication prior to and during study per fed and fasting status will presented by using the WHOdrug dictionary version 2021, the ACT classification name will be shown.

# 9. References

- Substance Abuse and Mental Health Services Administration. Key substance use and mental health indicators in the United States: Results from the 2018 National Survey on Drug Use and Health (HHS Publication No. PEP19-5068, NSDUH Series H-54). Rockville, MD: Center for Behavioral Health Statistics and Quality, Substance Abuse and Mental Health Services Administration; 2019.
- Substance Abuse and Mental Health Services Administration, Center for Behavioral Health Statistics and Quality. Treatment Episode Data Set (TEDS): 2005-2015. National Admissions to Substance Abuse Treatment Services. BHSIS Series S-91, HHS Publication No. (SMA) 17-5037. Rockville, MD: Substance Abuse and Mental Health Services Administration; 2017.
- Budney AJ, Higgins ST, Radonovich KJ, Novy PL. Adding voucher-based incentives to coping skills and motivational enhancement improves outcomes during treatment for marijuana dependence. J Consult Clin Psychol. 2000;68(6):1051-61. doi: 10.1037//0022-006x.68.6.1051.
- Budney AJ, Moore BA, Rocha HL, Higgins ST. Clinical trial of abstinence-based vouchers and cognitive-behavioral therapy for cannabis dependence. J Consult Clin Psychol. 2006;74(2):307-16. doi: 10.1037/0022-006x.4.2.307.
- Copeland J, Swift W, Roffman R, Stephens R. A randomized controlled trial of brief cognitive-behavioral interventions for cannabis use disorder. J Subst Abuse Treat. 2001;21(2):55-64; discussion 5-6. doi: 10.1016/s0740-5472(01)00179-9.
- 6. Stephens RS, Babor TF, Kadden R, Miller M. The Marijuana Treatment Project: rationale, design and participant characteristics. Addiction. 2002;97 Suppl 1:109-24. doi: 10.1046/j.1360-0443.97.s01.6.x.
- 7. Brezing CA, Levin FR. The Current State of Pharmacological Treatments for Cannabis Use Disorder and Withdrawal. Neuropsychopharmacology. 2018;43(1):173-94. doi: 10.1038/npp.2017.212.



| Study : 105 |
|------------------|
| Date : 19JAN2023 |

8. Weinstein AM, Gorelick DA. Pharmacological treatment of cannabis dependence. Curr Pharm Des. 2011;17(14):1351-8. doi: 10.2174/138161211796150846.

- 9. Aelis Farma. AEF0117 Investigator's Brochure. Edition 5.0; March 2022.
- 10. FDA. Guidance for Industry. Food-Effect Bioavailability and Fed Bioequivalence Studies. U.S. Department of Health and Human Services. U.S. Department of Health and HumanServices. Food and Drug Administration. Center for Drug Evaluation and Research (CDER). December 2002. Available from: <a href="https://www.fda.gov/files/drugs/published/Food-Effect-Bioavailability-and-Fed-Bioequivalence-Studies.pdf">https://www.fda.gov/files/drugs/published/Food-Effect-Bioavailability-and-Fed-Bioequivalence-Studies.pdf</a>.




Date: 19JAN2023

# 10. Tables to be presented in the report

# 10.1 Analysis sets

Table 1.1.1 Analysis sets - Subjects recruited

| | Total number of enrolled | | |
|---|---|---|---|
| | subjects | Fed | Fasting |
| | (n=xx) | (n=xx) | (n=xx) |
| Number of subjects in SAF | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of subjects excluded from SAF by reason for exclusion: | | | |
| Subjects who do not receive study medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of subjects in PK | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of subjects excluded from PK by reason for exclusion <sup>1</sup> : | | | |
| Subjects who do not receive study medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with plasma pharmacokinetic parameters not available | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects who vomited within 3 hours after dose administration | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Subjects with protocol deviations with significant influence on estimation of one or more PK parameter | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>1</sup>Subjects may present more than one reason.




Date: 19JAN2023

Table 1.1.2 Visits - SAF

| | | Total subjects Fed | | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Screening visit (Day -28 to -2) | n (%) | xx (xx.x%) | - | - |
| Baseline visit (Day -1) | n (%) | xx (xx.x%) | - | - |
| Day 1 | n (%) | xx (xx.x%) | - | - |
| Day 2 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 3 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 4 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 5 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 7 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 9 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 11 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Day 14 ±1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |




Date: 19JAN2023

Table 1.1.3 End of study - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Status of the subject | | | | |
| Completed | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Premature withdrawal n (%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Reason for premature<br>vithdrawal <sup>1</sup> | | | | |
| Total no-missing | n | xx | xx | xx |
| Screen failure | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol deviation | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawal by subject | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost to follow-up | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Study terminated by sponsor | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Technical problem | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | xx | XX |




Date: 19JAN2023

# 10.2 Descriptive analysis - SAF

# 10.2.1 Screening visit (Day -28 to -2)

Table 2.1.1 Demographic - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Age (years) | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx | XX |
| Weight (Kg) | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx | xx |
| Height (cm) | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx | xx |
| BMI (Kg/m²) | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |



Study: 105 Version: 1.0 Date: 19JAN2023

| | Total subjects | Fed | Fasting |
|---------|----------------|--------|---------|
| | (n=xx) | (n=xx) | (n=xx) |
| Missing | xx | xx | xx |




Date: 19JAN2023

Table 2.1.2 Sex, Ethnicity and Status - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Sex | | | | |
| Total no-missing | n | xx | xx | xx |
| Male | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Female | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | XX | xx |
| Ethnicity | | | | |
| Total no-missing | n | xx | xx | xx |
| Hispanic or Latino | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Hispanic or Latino | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Race | | | | |
| Total no-missing | n | xx | xx | xx |
| White | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Black or African | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| American | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Asian | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| American Indian or Alaska | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Native Hawaiian or other<br>Pacific islander | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | XX | XX |




Date : 19JAN2023

Table 2.1.3 Contraception - SAF

| | Table 2.1. | Total subjects Fed | | |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | Fasting<br>(n=xx) |
| Childbearing <sup>1</sup> | | ( | (**) | (=-7 |
| Ç | _ | | | |
| Total no-missing | n | xx | XX | XX |
| Fertile | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Post-menopausal | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Infertile / Sterile | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Pregnant or nursing female | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hysterectomy | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Annexectomy / Salpingectomy | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Tubal ligature / Tubal ligation | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ovariectomy | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | xx | xx |
| Contraception method <sup>2</sup> | | | | |
| Total no-missing | n | xx | xx | XX |
| Oral contraceptive | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Intra-uterine device | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Implant | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Diaphragm | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Condom with spermicide or jelly | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | xx | XX |

<sup>&</sup>lt;sup>1</sup>Only women.

<sup>&</sup>lt;sup>2</sup>Patients with child-bearing potential.




Date: 19JAN2023

# Table 2.1.4 Medical history - SAF

| | | Total aubicata End | | Fasting |
|------------------|-------|--------------------|------------|------------|
| | | Total subjects | Fed | |
| | | (n=xx) | (n=xx) | (n=xx) |
| Medical history | | | | |
| Total no-missing | n | xx | xx | xx |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Medical history | | | | |
| Total no-missing | n | XX | xx | xx |
| SOC 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |

The medical history will be presented by using the dictionary MedDRA version 25.0.




Date: 19JAN2023

Table 2.1.5 Ongoing medical history - SAF

| | | Total subjects | Fed | Fasting |
|-------------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| Ongoing medical history | | | | |
| Total no-missing | n | xx | xx | xx |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Ongoing medical history | | | | |
| Total no-missing | n | xx | xx | xx |
| SOC 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | XX | XX |

The ongoing medical history will be presented by using the dictionary MedDRA version 25.0.




Date: 19JAN2023

Table 2.1.6 Physical examination (Screening) - SAF

| | Total Subjects (n=xx) | | Fed<br>(n=xx) | | Fasting<br>(n=xx) | |
|---|---|---|---|---|---|---|
| | Total no-<br>missing | Normal | Total no-<br>missing | Normal | Total no-<br>missing | Normal |
| - | n | n (%) | n | n (%) | n | n (%) |
| Skin | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) |
| Head | xx | xx (xx.x%) | XX | xx (xx.x%) | xx | xx (xx.x%) |
| Eyes – Throat | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Thyroid | XX | xx (xx.x%) | XX | xx (xx.x%) | xx | xx (xx.x%) |
| Lungs | xx | xx (xx.x%) | XX | xx (xx.x%) | xx | xx (xx.x%) |
| Cardiovascular system | xx | xx (xx.x%) | XX | xx (xx.x%) | xx | xx (xx.x%) |
| Abdomen (Liver/spleen) | XX | xx (xx.x%) | XX | xx (xx.x%) | xx | xx (xx.x%) |
| Extremities | xx | xx (xx.x%) | XX | xx (xx.x%) | xx | xx (xx.x%) |
| Neurological | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) |




Date: 19JAN2023

Table 2.1.7 Vital signs (Screening) - SAF

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| Time between evaluation and visit Day 1 (days) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| Temperature (°C) | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | XX,XX | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | XX,XX | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| SBP - Supine (mmHg) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | XX,XX | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| DBP - Supine (mmHg) | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| Heart rate - Supine (bpm) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | xx,xx | xx |




Date: 19JAN2023

Table 2.1.8 Electrocardiogram (Normal/Abnormal) (Screening) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Electrocardiogram | | | | |
| Total no-missing | n | xx | xx | xx |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Does the result meet the definition of adverse event? | F | | | |
| Total no-missing | n | xx | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Does the result meet the definition of adverse event? (Any Yes per parameter)* | | | | |
| Total no-missing | n | xx | xx | xx |
| Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PR intervals | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| QT interval | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| QTcF interval | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | XX | XX |

<sup>\*</sup>More than one option per patient will be possible.




Date: 19JAN2023

Table 2.1.9 Electrocardiogram (Screening) - SAF

| | | Mean | Median | | |
|---|---|---|---|---|---|
| | n | (SD) | (Q1, Q3) | Min, Max | Missing |
| Time between ECG and dose (hours) | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Heart rate (BPM) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | XX |
| PR intervals (ms) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| QRS duration (ms) | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| QT interval (ms) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| QTcF Interval (ms) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |



Date: 19JAN2023

# Table 2.1.10 C-SSRS (Screening) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| C-SSRS | | | | |
| Total no-missing | n | xx | xx | xx |
| Suicidal Ideation or Behavior | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suicidal Ideation | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Wish to dead | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Non-specific active suicidal thoughts | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with any methods (not plan) without intent to act | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with some intent to act, without specific plan | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with specific plan and intent | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suicidal Behavior | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preparatory acts or behavior | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Aborted attempt | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Interrupted attempt | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Non-fatal suicide attempt | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Self-injorious behavior without suicidal intent | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |




Date: 19JAN2023

Table 2.1.11 Laboratory evaluation (Screening) - SAF

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| Time between evaluation and visit day 1 (days) | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |

Table 2.1.12 Percentage of numeric values and non-numeric values (Screening) - SAF

| | | Total subjects | Fed | Fasting |
|------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| Chemistry | | | | |
| Albumin (g/dl) | | | | |
| Total no-missing | n | xx | xx | xx |
| Numeric | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Value 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Hematology | | | | |
| Coagulation | | | | |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 




Date: 19JAN2023

# Table 2.1.13 Chemistry (Screening) - SAF

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|----------------|----|--------------|--------------------|----------|---------|
| Albumin (g/dL) | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |

ALT (GPT) (U/L)

...

AST (GOT) (U/L)

. . .

Carbon Dioxide (mmol/L)

. . .

Blood urea nitrogen (mg/dL)

- - -

Calcium (mg/dL)

- - -

Cholesterol Total (mg/dL)

• • •

Creatinine (mg/dL)

•••



Study: 105


Date: 19JAN2023

Mean Median (Q1, Q3) Min, Max n (SD) Missing CPK (U/L) Glucose (mg/dL) HDL (mg/dL) LDL (mg/dL) Phosphorus (mg/dL) Potassium (mmol/L) Sodium (mmol/L) Total Bilirubin (mg/dL) Total protein (g/dL) Triglycerides (mg/dL)



Study: 105


Date: 19JAN2023

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| Uric acid (mg/dL) | | | | | |
| FSH (mIU/mL) | | | | | |



Eosinophils (x10^3 µL)

### STATISTICAL ANALYSIS PLAN


Date: 19JAN2023

Table 2.1.14 Hematology (Screening) - SAF

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|----------------|----|--------------|--------------------|----------|---------|
| Hematocrit (%) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | XX |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |

# Hemoglobin (g/dL) MCV (fL) MCHC (g/L) Platelet count (x10^3 µL) RBC (x10<sup>6</sup> μL) WBC (x10<sup>3</sup> μL) Basophils (x10<sup>3</sup> µL)



Study : 105


Date : 19JAN2023

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| Lymphocytes (x10^3 µL) | | | | | |
| Monocytes (x10^3 μL) | | | | | |
| Neutrophils (x10^3 μL) | | | | | |




Date: 19JAN2023

# Table 2.1.15 Coagulation (Screening) - SAF

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|----------------|----|--------------|--------------------|----------|---------|
| INR | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |

## Prothrombine time (s)

- - -

## aPTT (s)

...




Date: 19JAN2023

# Table 2.1.16 Urinary analysis (Screening) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Color and appearance | | | | |
| Total no-missing | n | xx | xx | xx |
| Clear | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Cloudy | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hematuria | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | XX | XX |
| рН | n | xx | xx | |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx (xx.x%) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | xx (xx.x%) |
| | Missing | xx | xx | |
| Specific gravity | n | xx | xx | |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx (xx.x%) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | xx (xx.x%) |
| | Missing | xx | XX | |
| Glucose | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |




Date: 19JAN2023

| | | Total subjects | Fed | Fasting |
|------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | XX | xx |
| Protein | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | XX |
| Red blood cells | | | | |
| Total no-missing | n | xx | XX | XX |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| _eukocytes | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |




Date : 19JAN2023

| | | Total subjects | Fed | Fasting |
|------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | XX | xx |
| Ketones | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | XX | xx |
| Bilirubin | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |




Date: 19JAN2023

| | | Total subjects | Fed | Fasting |
|------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| Urobilinogen | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Vitrite | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |




Date: 19JAN2023

# 10.2.2 Baseline (Day -1)

Table 2.2.1 Weight and BMI (Baseline) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Weight (Kg) | N | xx | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx | xx |
| BMI (Kg/m²) | N | XX | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx | xx |



Study : 105


Date: 19JAN2023

Table 2.2.2 Physical examination (Baseline) - SAF

| | | Total Subjects (n=xx) | | Fed<br>(n=xx) | | eting<br>=xx) |
|---|---|---|---|---|---|---|
| | Total no-<br>missing | Normal | Total no-<br>missing | Normal | Total no-<br>missing | Normal |
| | n | n (%) | n | n (%) | n | n (%) |
| Skin | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Head | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Eyes and Throat | xx | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) |
| Thyroid | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Lungs | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Cardiovascular system | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Abdomen (Liver/spleen) | xx | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) |
| Extremities | xx | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) |
| Neurological | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |




Date : 19JAN2023

Table 2.2.3 Vital signs (Baseline) - SAF

| | N | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| Time between evaluation and visit day 1 (days) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Temperature (°C) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| SBP - Supine (mmHg) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| DBP - Supine (mmHg) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Heart rate - Supine (bpm) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |




Date: 19JAN2023

Table 2.2.4 Electrocardiogram (Normal/Abnormal) (Baseline) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Electrocardiogram | | | | |
| Total no-missing | n | xx | xx | xx |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Does the result meet the definition adverse event? | ı of | | | |
| Total no-missing | n | xx | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Does the result meet the definition adverse event? (Any Yes parameter)* | of<br>per | | | |
| Total no-missing | n | xx | xx | xx |
| Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PR intervals | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| QT interval | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| QTcF interval | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | XX | XX |

<sup>\*</sup>More than one option per patient will be possible




Date: 19JAN2023

Table 2.2.5 Electrocardiogram (Baseline) - SAF

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| Time between ECG and dose (hours) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Heart rate (BPM) | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| PR intervals (ms) | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| QRS duration (ms) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| QT interval (ms) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| QTcF interval (ms) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |




Date: 19JAN2023

# Table 2.2.6 C-SSRS (Baseline) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| C-SSRS | | (n=xx) | (n=xx) | (n=xx) |
| Total no-missing | n | xx | xx | xx |
| Suicidal Ideation or Behavior | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suicidal Ideation | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Wish to dead | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Non-specific active suicidal thoughts | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with any methods (not plan) without intent to act | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with some intent to act, without specific plan | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with specific plan and intent | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suicidal Behavior | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preparatory acts or behavior | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Aborted attempt | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Interrupted attempt | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Non-fatal suicide attempt | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Self-injorious behavior without suicidal intent | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |




Date: 19JAN2023

Table 2.2.7 Laboratory evaluation (Baseline) - SAF

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| Time between evaluation and visit day 1 (days) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | XX |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |

Table 2.2.8 Percentage of numeric and non-numeric values (Baseline) - SAF

| | | Total subjects | Fed | Fasting |
|------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| Chemistry | | | | |
| Albumin (g/dl) | | | | |
| Total no-missing | n | xx | xx | xx |
| Numeric | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Value 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Hematology | | | | |
| Coagulation | | | | |




Date: 19JAN2023

# Table 2.2.9 Chemistry (Baseline) - SAF

| | | Mean | Median | | |
|----------------|----|-------------|------------|----------|---------|
| | n | (SD) | (Q1, Q3) | Min, Max | Missing |
| Albumin (g/dL) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | XX |

ALP (U/L)

...

ALT (GPT) (U/L)

...

AST (GOT) (U/L)

. . .

Bicarbonate (mEq(L)

. . .

Blood urea nitrogen (mg/dL)

Calcium (mg/dL)

- - -

Cholesterol Total (mg/dL)

• • •

Creatinine (mg/dL)

• • •



Study : 105


Date : 19JAN2023

Mean Median n (SD) (Q1, Q3) Min, Max Missing

| CPK (U/L) |
|-------------------------|
| Glucose (mg/dL) |
| <del></del> |
| HDL (mg/dL) |
| LDL (mg/dL) |
| Phosphorus (mg/dL) |
| Potassium (mmol/L) |
| <del></del> |
| Sodium (mmol/L) |
| Total Bilirubin (mg/dL) |
| Total protein (g/dL) |
| Triglycerides (mg/dL) |
| rraivcerraes (Ma/aL) |



Study: 105


Date: 19JAN2023

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| Uric acid (mg/dL) | | | | | |




Date: 19JAN2023

# Table 2.2.10 Hematology (Baseline) - SAF

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|----------------|----|--------------|--------------------|----------|---------|
| Hematocrit (%) | | | | | |
| Total subjects | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | XX |

# Hemoglobin (g/dL) MCV (fL) MCHC (g/L) Platelet count (x10^3 µL) RBC (x10<sup>6</sup> μL) WBC (x10<sup>3</sup> μL) Basophils (x10<sup>3</sup> µL)

Eosinophils (x10<sup>3</sup> μL)

• • •



Study : 105


Date : 19JAN2023

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| Lymphocytes (x10^3 µL) | | | | | |
| Monocytes (x10^3 μL) | | | | | |
| Neutrophils (x10^3 μL) | | | | | |




Date: 19JAN2023

# Table 2.2.11 Coagulation (Baseline) - SAF

| | n | Mean<br>(SD) | Median<br>(Q1, Q3) | Min, Max | Missing |
|----------------|----|--------------|--------------------|----------|---------|
| INR | | | | | |
| Total subjects | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fed | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | xx (xx,xx) | (xx,xx) | xx |

## Prothrombine time (s)

...

## aPTT (s)

...




Date: 19JAN2023

# Table 2.2.12 Urinary analysis (Baseline) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Color and appearance | | | | |
| Total no-missing | n | xx | xx | xx |
| Limpid | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Cloudy | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hematuria | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| рН | n | xx | xx | |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx (xx.x%) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | xx (xx.x%) |
| | Missing | xx | xx | |
| Specific gravity | n | xx | xx | |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx (xx.x%) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | xx (xx.x%) |
| | Missing | xx | xx | |
| Glucose | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |




Date: 19JAN2023

| | | Total subjects | Fed | Fasting |
|------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | XX | xx |
| rotein rotein | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | XX | xx |
| Red blood cells | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | XX |
| eukocytes | | | | |
| Total no-missing | n | XX | xx | XX |



Study : 105


Date: 19JAN2023

| | | Total subjects | Fed | Fasting |
|------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | XX | xx |
| Ketones | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | xx | xx |
| Bilirubin | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |



Study : 105


Date: 19JAN2023

| | | Total subjects | Fed | Fasting |
|------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| Missing | n | xx | xx | xx |
| Jrobilinogen | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| litrite | | | | |
| Total no-missing | n | xx | xx | xx |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Trace | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3+ | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |




Date: 19JAN2023

# 10.2.3 Follow-up

Table 2.3.1 CRU discharge (24 hours) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Was the subject experiencing any | | | | |
| adverse event at the scheduled time | | | | |
| of the CRU discharge? | | | | |
| Total no-missing | n | xx | xx | xx |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Was the subject discharged from CRU as scheduled? Total no-missing | n | xx | xx | xx |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| Reason¹ | | | | |
| Total no-missing | n | xx | xx | xx |
| Adverse Event | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | XX |




Date: 19JAN2023

# Table 2.3.2 Tests (days 3,4,5,7,9,11) - SAF

| | | Total subjects | Fed | Fasting |
|---------------------|-------|----------------|------------|------------|
| | | (n=xx) | (n=xx) | (n=xx) |
| Alcohol breath test | | | | |
| Total no-missing | n | xx | xx | xx |
| Any test Positive | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| All Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |

# All Negative n (%) xx (xx.x%) xx (xx.x%) xx (xx.x%) Missing n xx xx xx xx xx Amphetamine test ... Benzodiazepines test ... Cannabinoids test ... Cocaine (metabolite) test ...

## Methamphetamine test

...

## Methadone test



Study: 105


Date: 19JAN2023

Total subjects Fed Fasting

(n=xx) (n=xx) (n=xx)

Table 2.3.3 Weight and BMI (312 h) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Weight (Kg) | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx | xx |
| BMI (Kg/m²) | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx | xx |

Table 2.3.4 Pregnancy test (312 hours) - SAF

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Pregnancy test result <sup>1</sup> | | | | |
| Total no-missing | n | XX | xx | xx |
| Positive | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | XX |



Study : 105


Date: 19JAN2023

# 10.3 Primary objective

## 10.3.1 Pharmacokinetic endpoints

Table 3.1.1 Descriptive analysis of pharmacokinetic endpoints - PK

| | n | Mean<br>(SD) | Geometric<br>mean | cv | Median<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|---|---|
| C <sub>max</sub> (ng/mL) | | | | | | | |
| Fed | xx | xx.x (xx.x) | XX.X | XX.X | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | xx.x | XX.X | xx (xx,xx) | (xx,xx) | xx |
| T <sub>max</sub> (hours) | | | | | | | |
| Fed | XX | - | - | - | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | - | - | - | xx (xx,xx) | (xx,xx) | xx |
| t <sub>lag</sub> (hours) | | | | | | | |
| Fed | xx | - | - | - | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | - | - | - | xx (xx,xx) | (xx,xx) | xx |
| AUC <sub>0-t</sub> (hours*ng/mL) | | | | | | | |
| Fed | xx | xx.x (xx.x) | xx.x | XX.X | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | XX.X | XX.X | xx (xx,xx) | (xx,xx) | xx |
| AUC₀<br>(hours*ng/mL) | | | | | | | |
| Fed | XX | xx.x (xx.x) | XX.X | XX.X | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | XX.X | XX.X | xx (xx,xx) | (xx,xx) | xx |




Date: 19JAN2023

# Table 3.1.2 Regression analysis of pharmacokinetic endpoints - PK

| | State effect<br>p-value | Geometric Mean ratio<br>CI 90% |
|---|---|---|
| C <sub>max</sub> (ng/mL) | x.xxxx | xx.x (xx.x, xx.x) |
| AUC <sub>0-t</sub> (hours*ng/mL) | x.xxxx | xx.x (xx.x, xx.x) |
| AUC <sub>0-∞</sub> (hours*ng/mL) | x.xxxx | xx.x (xx.x, xx.x) |



Study : 105

Date: 19JAN2023

# 10.4 Secondary objectives

# 10.4.1 Pharmacokinetic secondary endpoints

Table 4.1.1 Descriptive analysis of pharmacokinetic secondary endpoints - PK

| | | Mean | Geometric | Median | | | |
|---|---|---|---|---|---|---|---|
| | n | (SD) | mean | CV | (Q1, Q3) | Min, Max | Missing |
| AUC <sub>extrap</sub> (%) | | | | | | | |
| Fed | xx | xx.x (xx.x) | XX.X | xx.x | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | XX.X | xx.x | xx (xx,xx) | (xx,xx) | xx |
| C <sub>24h</sub> (ng/mL) | | | | | | | |
| Fed | xx | xx.x (xx.x) | XX.X | xx.x | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | XX.X | xx.x | xx (xx,xx) | (xx,xx) | xx |
| t <sub>1/2</sub> (hours) | | | | | | | |
| Fed | XX | - | - | - | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | - | - | - | xx (xx,xx) | (xx,xx) | xx |
| CL/F (L/hours) | | | | | | | |
| Fed | xx | xx.x (xx.x) | XX.X | xx.x | xx (xx,xx) | (xx,xx) | xx |
| Fasting | XX | xx.x (xx.x) | XX.X | xx.x | xx (xx,xx) | (xx,xx) | xx |
| Vd/F (L) | | | | | | | |
| Fed | XX | xx.x (xx.x) | XX.X | xx.x | xx (xx,xx) | (xx,xx) | xx |
| Fasting | xx | xx.x (xx.x) | XX.X | XX.X | xx (xx,xx) | (xx,xx) | xx |




Date: 19JAN2023

# 10.4.2 Safety endpoints - Adverse Events

Table 4.2.1 General summary of adverse events – SAF

| | | ed<br>exx) | Fasting<br>(n=xx) | |
|---|---|---|---|---|
| | Number of subjects | Number of events | Number of subjects | Number of events |
| | n (%) | E | n (%) | E |
| Any AE | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Any related AE | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Any serious AE | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Any serious related AE | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Any AE: | | | | |
| Severity | | | | |
| Mild | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Moderate | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Severe | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Outcome | | | | |
| Recovered/Resolved | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Recovering/Resolving | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Not recovered/Not resolved | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Recovered/Resolved with sequelae | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Fatal | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Unknown | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Action taken with study treatment | | | | |
| Dose not changed | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Drug withdrawn | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Drug interrupted | xx (xx.x%) | xx | xx (xx.x%) | xx |



Date: 19JAN2023

| | | ed<br>xx) | | ting<br>:xx) |
|---|---|---|---|---|
| | Number of subjects | | | Number of events |
| | n (%) | E | n (%) | E |
| Dose increased | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Dose reduced | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Not applicable | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Unknown | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Related with alternative causality or confounding factors | | | | |
| Yes | xx (xx.x%) | xx | xx (xx.x%) | xx |
| No | xx (xx.x%) | xx | xx (xx.x%) | XX |



Study: 105

Date: 19JAN2023

Table 4.2.2 AE I (Fed) - SAF

| | | | | | Severity | | Causa | lity | Related with altern | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Duration | · | | | | | · | |
| | Nº pat. (%) | Nº AE | (minutes)* | Mild | Moderate | Severe | Not Related | Related | Yes | No |
| Overall | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| ••• | | | | | | | | | | |
| SOC 2 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | XX | xx |

\*Mean(SD)

The AE will be presented by using the MedDRA dictionary version 25.0.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 



Study : 105

Date: 19JAN2023


Table 4.2.3 AE II (Fed) - SAF

| | TUDIO TILIO TE II (I OU) | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Action / | Study treatm | nent | | | | | Outcome | | | |
| | Nº pat. | Nº | Dose not | Drug | Drug | Dose | Dose | Not | | Recovered / | Recovering / | Not recovered | With | | |
| - | (%) | ΑE | changed | withdrawn | interrupted | increased | reduced | applicable | Unknown | Resolved | Resolving | / Not resolved | sequelae | Fatal | Unknown |
| <u>Overall</u> | xx (xx.x) | xx | xx | xx | XX | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | xx | xx | xx | xx | XX | xx | xx | xx | xx | xx | XX | xx | xx |
| PT 1 | xx (xx.x) | XX | XX | xx | xx | XX | xx | XX | XX | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | XX | xx | xx | XX | xx | XX | xx | xx | xx | xx | xx | xx | XX |
| SOC 2 | xx (xx.x) | XX | XX | xx | xx | XX | xx | XX | XX | xx | xx | xx | xx | xx | XX |
| PT 1 | xx (xx.x) | XX | XX | xx | xx | XX | xx | XX | XX | xx | xx | xx | xx | xx | XX |
| PT 2 | xx (xx.x) | XX | XX | xx | xx | XX | xx | XX | xx | xx | xx | xx | xx | xx | XX |

The AE will be presented by using the MedDRA dictionary version 25.0.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 



Study : 105 Version : 1.0

Date: 19JAN2023

Table 4.2.4 AE III (Fed) - SAF

| | | | Ser | ious | | | Serious | criteria | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Nº pat. (%) | Nº AE | No | Yes | Death | Hospitalization<br>or<br>prolongation<br>of existing<br>hospitalization | Congenital<br>anomaly or<br>birth defect | Other<br>medically<br>important<br>event | Life<br>threatening | Significant<br>disability /<br>incapacity |
| <u>Overall</u> | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| SOC 2 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| ••• | | | | | | | | | | |

The AE will be presented by using the MedDRA dictionary version 25.0.



| Study : 105 |
|------------------|
| Date : 19IAN2023 |

Table 4.2.5 AE I (Fasting) - SAF Table 4.2.6 AE II (Fasting) - SAF Table 4.2.7 AE III (Fasting) - SAF




Date: 19JAN2023

# 10.4.3 Safety endpoints - Treatment Emergent Adverse Events

Table 4.3.1 General summary of treatment emergent adverse events – SAF

| | | ed<br>xxx) | | eting<br>exx) |
|---|---|---|---|---|
| | Number of subjects | Number of events | Number of subjects | Number of events |
| | n (%) | E | n (%) | E |
| Any TEAE | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Any related TEAE | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Any serious TEAE | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Any serious related TEAE | xx (xx.x%) | XX | xx (xx.x%) | xx |
| Any TEAE: | | | | |
| Severity | | | | |
| Mild | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Moderate | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Severe | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Outcome | | | | |
| Recovered/Resolved | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Recovering/Resolving | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Not recovered/Not resolved | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Recovered/Resolved with sequelae | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Fatal | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Unknown | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Action taken with study treatment | | | | |
| Dose not changed | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Drug withdrawn | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Drug interrupted | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Dose increased | xx (xx.x%) | xx | xx (xx.x%) | xx |



Study : 105


Date: 19JAN2023

| | | ed<br>exx) | | ting<br>:xx) |
|---|---|---|---|---|
| | Number of subjects | Number of events | Number of subjects | Number of events |
| | n (%) | E | n (%) | n (%) E |
| Dose reduced | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Not applicable | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Unknown | xx (xx.x%) | xx | xx (xx.x%) | xx |
| Related with alternative causality or confounding factors | | | | |
| Yes | xx (xx.x%) | xx | xx (xx.x%) | xx |
| No | xx (xx.x%) | xx | xx (xx.x%) | XX |



Study : 105


Date : 19JAN2023

Table 4.3.2 TEAE I (Fed) - SAF

| | | | | | Severity | | Causa | lity | Related with altern | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Duration | | | | | | | |
| | Nº pat. (%) | Nº TEAE | (minutes)* | Mild | Moderate | Severe | Not Related | Related | Yes | No |
| <u>Overall</u> | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| SOC 2 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |

<sup>\*</sup>Mean(SD)

The TEAE will be presented by using the MedDRA dictionary version 25.0.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 



Study: 105

Date: 19JAN2023

Table 4.3.3 TEAE II (Fed) - SAF

| | | | | | Action / | Study treatm | nent | | | Outcome | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Nº pat. | Nº | Dose not | Drug | Drug | Dose | Dose | Not | | Recovered / | Recovering / | Not recovered | With | | |
| | (%) | TEAE | changed | withdrawn | interrupted | increased | reduced | applicable | Unknown | Resolved | Resolving | / Not resolved | sequelae | Fatal | Unknown |
| <u>Overall</u> | xx (xx.x) | xx | XX | xx | xx | XX | xx | XX | xx | xx | xx | xx | xx | xx | xx |
| SOC 1 | xx (xx.x) | XX | XX | xx | xx | XX | xx | XX | XX | xx | xx | xx | XX | xx | xx |
| PT 1 | xx (xx.x) | XX | XX | xx | xx | XX | xx | XX | XX | xx | xx | xx | XX | xx | xx |
| PT 2 | xx (xx.x) | XX | XX | xx | xx | XX | xx | XX | XX | xx | xx | xx | XX | xx | xx |
| *** | | | | | | | | | | | | | | | |
| SOC 2 | xx (xx.x) | xx | XX | xx | xx | XX | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |

The TEAE will be presented by using the MedDRA dictionary version 25.0.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 



Study: 105

Date: 19JAN2023

Table 4.3.4 TEAE III (Fed) - SAF

| | | | Ser | ious | | | Serious | criteria | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N° pat. (%) | Nº TEAE | No | Yes | Death | Hospitalization<br>or<br>prolongation<br>of existing<br>hospitalization | Congenital<br>anomaly or<br>birth defect | Other<br>medically<br>important<br>event | Life<br>threatening | Significant<br>disability /<br>incapacity |
| <u>Overall</u> | xx (xx.x) | xx | xx | xx | xx | XX | xx | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| ••• | | | | | | | | | | |
| SOC 2 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | xx | XX | xx | xx | xx | xx |
| ••• | | | | | | | | | | |

The TEAE will be presented by using the MedDRA dictionary version 25.0.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 



Study: 105

Date: 19JAN2023

Table 4.3.5 TEAE III (Fed) - SAF

| | | | Seri | ous | | | Serious | criteria | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Nº pat. (%) | Nº TEAE | Yes | No | Death | Hospitalization<br>or<br>prolongation<br>of existing<br>hospitalization | Congenital<br>anomaly or<br>birth defect | Other<br>medically<br>important<br>event | Life<br>threatening | Significant<br>disability /<br>incapacity |
| <u>Overall</u> | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| SOC 2 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx |

The TEAE will be presented by using the MedDRA dictionary version 25.0.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 



| Study : 105 |
|------------------|
| Date : 19JAN2023 |

Table 4.3.6 TEAE I (Fasting) - SAF Table 4.3.7 TEAE II (Fasting) - SAF Table 4.3.8 TEAE III (Fasting) - SAF




Date: 19JAN2023

# 10.4.4 Safety endpoints - Vital Signs

Table 4.4.1 Time between evaluation and dose (hours) - SAF

| | | Fed | Fasting |
|----------|----------------|-------------------|-------------------|
| | | (n=xx) | (n=xx) |
| Pre-dose | n | XX | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | XX |
| 1 hour | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 2 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 4 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 8 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |




Date: 19JAN2023

| | | Fed<br>(n=xx) | Fasting<br>(n=xx) |
|-----------|----------------|-------------------|-------------------|
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 11 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 24 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 48 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 240 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 312 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |



| Study : 105 |
|-----------------|
| Date: 19JAN2023 |

| | Fed | Fasting |
|---------|--------|---------|
| | (n=xx) | (n=xx) |
| Missing | xx | xx |

For the heart rate and blood pressure variables same table format as Table 4.4.1:

Table 4.4.2 SBP - Supine (mmHg) - SAF Table 4.4.3 DBP - Supine (mmHg) - SAF Table 4.4.4 Heart rate - Supine (bpm) - SAF

Table 4.4.5 Oral temperature (°C) - SAF

| | | Fed | Fasting |
|-----------|----------------|-------------------|-------------------|
| | | (n=xx) | (n=xx) |
| Baseline | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | XX |
| 24 hours | n | xx | XX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | XX |
| 312 hours | n | xx | XX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |




Date: 19JAN2023

# 10.4.5 Safety endpoints - Electrocardiogram

Table 4.5.1 Electrocardiogram (Normal/Abnormal) - SAF

| l able 4 | 1.5.1 Electrocardiogram (N | (Normal/Abhormal) - SAF | |
|---|---|---|---|
| | | Fed | Fasting |
| | | (n=xx) | (n=xx) |
| Electrocardiogram (pre-dose) | | | |
| Total no-missing | n | xx | xx |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the day | definition of | | |
| Total no-missing | n | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the dadverse event? (Any Yes per part | | | |
| Total no-missing | n | xx | xx |
| Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) |
| PR intervals | n (%) | xx (xx.x%) | xx (xx.x%) |
| QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) |
| QT interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QTcF interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Electrocardiogram (1 hour) | | | |
| Total no-missing | n | xx | xx |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |




Date: 19JAN2023

| | | Fed | Fasting |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Missing | n | xx | xx |
| Does the result meet the dadverse event? | definition of | | |
| Total no-missing | n | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the dadverse event? (Any Yes per par | | | |
| Total no-missing | n | xx | xx |
| Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) |
| PR intervals | n (%) | xx (xx.x%) | xx (xx.x%) |
| QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) |
| QT interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QTcF interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Electrocardiogram (2 hours) | | | |
| Total no-missing | n | xx | xx |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the dadverse event? | definition of | | |
| Total no-missing | n | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |




Date : 19JAN2023

| Total no-missing n xx xx All Normal n (%) xx (xx.x%) xx (xx.x%) Any Abnormal n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx xx Does the result meet the definition of adverse event? Total no-missing n xx xx xx | | | Fed | Fasting |
|---|---|---|---|---|
| Adverse event? (Any Yes per parameter)* Total no-missing n | | | (n=xx) | (n=xx) |
| Total no-missing | Does the result meet the c | definition of | | |
| Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) QT interval n (%) xx (xx.x%) xx (xx.x%) QT or intervals n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Electrocardiogram (4 hours) xx xx xx Total no-missing n xx (xx.x%) xx (xx.x%) All Normal n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Does the result meet the definition of odverse event? xx xx xx Total no-missing n xx xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Obes the result meet the definition of odverse event? (Any Yes per parameter)* xx xx Total no-missing n xx xx Total no-missing n xx xx A | adverse event? (Any Yes per par | rameter)* | | |
| PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) QT interval n (%) xx (xx.x%) xx (xx.x%) QT of intervals n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Electrocardiogram (4 hours) xx xx xx Total no-missing n xx (xx.x%) xx (xx.x%) All Normal n (%) xx (xx.x%) xx (xx.x%) Any Abnormal n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Does the result meet the definition of adverse event? xx (xx.x%) xx (xx.x%) Total no-missing n xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Oces the result meet the definition of adverse event? (Any Yes per parameter)* xx xx Total no-missing n xx xx Does the result meet the definition of adverse event? (Any Yes per parameter)* xx xx | Total no-missing | n | xx | xx |
| QRS duration n (%) xx (xx.x%) xx (xx.x%) QT interval n (%) xx (xx.x%) xx (xx.x%) QTcF intervals n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Electrocardiogram (4 hours) xx xx xx Total no-missing n xx (xx.x%) xx (xx.x%) All Normal n (%) xx (xx.x%) xx (xx.x%) Any Abnormal n (%) xx (xx.x%) xx (xx.x%) Does the result meet the definition of adverse event? n (%) xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx xx Does the result meet the definition of adverse event? (Any Yes per parameter)* xx xx xx Total no-missing n xx xx xx Does the result meet the definition of adverse event? (Any Yes per parameter)* xx xx Total no-missing < | Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) |
| QT interval n (%) xx (xx.x%) xx (xx.x%) QTcF intervals n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Electrocardiogram (4 hours) xx xx xx Total no-missing n xx (xx.x%) xx (xx.x%) Any Abnormal n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Does the result meet the definition of adverse event? n (%) xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Obes the result meet the definition of adverse event? (Any Yes per parameter)* xx xx Total no-missing n xx xx Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | PR interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QTcF intervals n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Electrocardiogram (4 hours) Total no-missing n xx xx All Normal n (%) xx (xx.x%) xx (xx.x%) Any Abnormal n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Does the result meet the definition of adverse event? n (%) xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Does the result meet the definition of adverse event? (Any Yes per parameter)* xx xx Total no-missing n xx xx Total no-missing n xx xx Total no-missing n xx xx PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing n xx xx Electrocardiogram (4 hours) n xx xx Total no-missing n xx (xx.x%) xx (xx.x%) All Normal n (%) xx (xx.x%) xx (xx.x%) Any Abnormal n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Does the result meet the definition of olderse event? n (%) xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Missing n xx (xx.x%) xx (xx.x%) Obes the result meet the definition of olderse event? (Any Yes per parameter)* xx xx Total no-missing n xx xx Does the result meet the definition of olderse event? (Any Yes per parameter)* xx xx Total no-missing n xx xx Does the result meet the definition of olderse event? (Any Yes per parameter)* xx xx Total no-missing n xx xx Does the result meet the definition of olderse event? (Any Yes per parameter)* xx <td>QT interval</td> <td>n (%)</td> <td>xx (xx.x%)</td> <td>xx (xx.x%)</td> | QT interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| Electrocardiogram (4 hours) Total no-missing n n xx xx xx All Normal n (%) xx (xx.x%) xx (xx.x%) Any Abnormal n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx xx Obes the result meet the definition of adverse event? Total no-missing n xx xx xx Any Yes n (%) xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx xx Any Yes n (%) xx (xx.x%) xx (xx.x%) Obes the result meet the definition of adverse event? (Any Yes per parameter)* Total no-missing n xx xx xx Does the result meet the definition of adverse event? (Any Yes per parameter)* Total no-missing n xx xx xx Heart rate n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) Ax (xx.x%) xx (xx.x%) | QTcF intervals | n (%) | xx (xx.x%) | xx (xx.x%) |
| Total no-missing n | Missing | n | xx | xx |
| All Normal | Electrocardiogram (4 hours) | | | |
| Any Abnormal n (%) | Total no-missing | n | xx | xx |
| Missing n xx xx Does the result meet the definition of adverse event? n xx xx Total no-missing n xx (xx.x%) xx (xx.x%) Any Yes n (%) xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Does the result meet the definition of adverse event? (Any Yes per parameter)* xx xx Total no-missing n xx xx Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | All Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Does the result meet the definition of adverse event? n xx xx Total no-missing n xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx Does the result meet the definition of adverse event? (Any Yes per parameter)* n xx xx Total no-missing n xx xx xx Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Total no-missing n xx xx xx Any Yes n (%) xx (xx.x%) xx (xx.x%) All No n (%) xx (xx.x%) xx (xx.x%) Missing n xx xx xx Oces the result meet the definition of adverse event? (Any Yes per parameter)* Total no-missing n xx xx xx Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | Missing | n | xx | xx |
| Total no-missing n | Does the result meet the c | definition of | | |
| Any Yes | adverse event? | | | |
| All No | Total no-missing | n | xx | xx |
| Missing n xx xx Does the result meet the definition of adverse event? (Any Yes per parameter)* Total no-missing n xx xx Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) |
| Does the result meet the definition of adverse event? (Any Yes per parameter)* Total no-missing n xx xx Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | All No | n (%) | xx (xx.x%) | xx (xx.x%) |
| adverse event? (Any Yes per parameter)* Total no-missing n xx xx Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | Missing | n | xx | xx |
| Total no-missing n xx xx Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | Does the result meet the o | definition of | | |
| Heart rate n (%) xx (xx.x%) xx (xx.x%) PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | adverse event? (Any Yes per par | rameter)* | | |
| PR interval n (%) xx (xx.x%) xx (xx.x%) QRS duration n (%) xx (xx.x%) xx (xx.x%) | Total no-missing | n | xx | xx |
| QRS duration n (%) xx (xx.x%) xx (xx.x%) | Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) |
| | PR interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QT interval n (%) xx (xx.x%) xx (xx.x%) | QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) |
| | QT interval | n (%) | xx (xx.x%) | xx (xx.x%) |



Study : 105


Date: 19JAN2023

| | | Fed | Fasting |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| QTcF intervals | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | XX |
| Electrocardiogram (8 hours) | | | |
| Total no-missing | n | xx | XX |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the defined verse event? | nition of | | |
| Total no-missing | n | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the definational definition of the definition | | | |
| Total no-missing | n | xx | xx |
| Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) |
| PR interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) |
| QT interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QTcF intervals | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Electrocardiogram (11 hours) | | | |
| Total no-missing | n | xx | xx |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |




Date: 19JAN2023

| | | Fed | Fasting |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Does the result meet the deadverse event? | efinition of | | |
| Total no-missing | n | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the deadverse event? (Any Yes per para | | | |
| Total no-missing | n | xx | xx |
| Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) |
| PR interval | n (%) | xx (xx.x%) | xx (xx.x% |
| QRS duration | n (%) | xx (xx.x%) | xx (xx.x% |
| QT interval | n (%) | xx (xx.x%) | xx (xx.x% |
| QTcF intervals | n (%) | xx (xx.x%) | xx (xx.x% |
| Missing | n | xx | xx |
| Electrocardiogram (24 hours) | | | |
| Total no-missing | n | xx | xx |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x% |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x% |
| Missing | n | xx | xx |
| Does the result meet the deadverse event? | efinition of | | |
| Total no-missing | n | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x% |
| Missing | n | xx | xx |

Does the result meet the definition of adverse event? (Any Yes per parameter)\*




Date: 19JAN2023

| | | Fed | Fasting |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Total no-missing | n | xx | XX |
| Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) |
| PR interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) |
| QT interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QTcF intervals | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | XX |
| Electrocardiogram (240 hours) | | | |
| Total no-missing | n | xx | xx |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the definition adverse event? | on of | | |
| Total no-missing | n | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the definition adverse event? (Any Yes per parameter | | | |
| Total no-missing | n | xx | xx |
| Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) |
| PR interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) |
| QT interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QTcF intervals | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |



Study : 105


Date: 19JAN2023

| | | Fed | Fasting |
|-------------------------------|---------------|------------|------------|
| | | (n=xx) | (n=xx) |
| Electrocardiogram (312 hours) | | | |
| Total no-missing | n | xx | xx |
| All Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Any Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the o | definition of | | |
| Total no-missing | n | xx | xx |
| Any Yes | n (%) | xx (xx.x%) | xx (xx.x%) |
| All No | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| Does the result meet the o | | | |
| Total no-missing | n | xx | xx |
| Heart rate | n (%) | xx (xx.x%) | xx (xx.x%) |
| PR interval | n (%) | xx (xx.x%) | xx (xx.x% |
| QRS duration | n (%) | xx (xx.x%) | xx (xx.x%) |
| QT interval | n (%) | xx (xx.x%) | xx (xx.x%) |
| QTcF intervals | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | XX |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

\*More than one option per subject will be possible.




Date: 19JAN2023

# Table 4.5.2 Time between ECG and dose (hours) - SAF

| | | Fed<br>(n=xx) | Fasting<br>(n=xx) |
|---------|----------------|-------------------|-------------------|
| re-dose | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| hour | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | XX |
| hours | n | xx | XX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | XX | xx |




Date: 19JAN2023

| | | Fed | Fasting |
|-----------|----------------|-------------------|-------------------|
| | | (n=xx) | (n=xx) |
| 1 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | XX |
| 24 hours | n | xx | XX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 240 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 312 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | XX | xx |

For the rest of ECG parameters same table format as table 5.3.2

Table 4.5.3 Heart rate (BPM) - SAF Table 4.5.4 PR intervals (ms) - SAF Table 4.5.5 QRS duration (ms) - SAF Table 4.5.6 QT interval (ms) - SAF Table 4.5.7 QTcF interval (ms) - SAF



Study : 105


Date: 19JAN2023

# 10.5 Safety analysis

## 10.5.1 Laboratory parameters - SAF

Table 5.1.1 Time between evaluation and dose (days) - SAF

| | | Fed | Fasting |
|-------------------|----------------|-------------------|------------------|
| | | (n=xx) | (n=xx) |
| Baseline (Day -1) | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 4 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 312 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x |
| | Missing | xx | xx |



Study: 105


Date: 19JAN2023

## Table 5.1.2 Non numeric values - SAF

| | | Base | eline | 24 h | ours | 312 hours | |
|---|---|---|---|---|---|---|---|
| | | Fed | Fasting | Fed | Fasting | Fed | Fasting |
| | | (n=xx) | (n=xx) | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Chemistry | | | | | | | |
| Albumin (g/dl) | | | | | | | |
| Total no-missing | n | xx | xx | xx | xx | xx | xx |
| Numeric | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Value 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx | xx | xx | xx |
| ••• | | | | | | | |
| Hematology | | | | | | | |
| ••• | | | | | | | |
| Coagulation | | | | | | | |



Study : 105

Date: 19JAN2023

Table 5.1.3 Chemistry - Albumin (g/dl) - SAF

| | | Fed<br>(n=xx) | Fasting<br>(n=xx) |
|-------------------|----------------|-------------------|-------------------|
| Baseline (Day -1) | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 24 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 312 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |

For the rest of chemistry, hematology and coagulation parameters same table format as table 5.1.3:

Table 5.1.4 Chemistry – ALP (U/L) - SAF
Table 5.1.5 Chemistry - ALT (GPT) (U/L) - SAF
Table 5.1.6 Chemistry - AST (GOT) (U/L) – SAF
Table 5.1.7 Chemistry – Bicarbonate (mEq/L) - SAF
Table 5.1.8 Chemistry – Blood urea nitrogen (mg/dL) - SAF
Table 5.1.9 Chemistry - Calcium (mg/dL) - SAF
Table 5.1.10 Chemistry - Total Cholesterol (mg/dL) – SAF
Table 5.1.11 Chemistry - Creatinine (mg/dL) – SAF
Table 5.1.12 Chemistry - CPK (U/L) – SAF
Table 5.1.13 Chemistry - Glucose (mg/dL) - SAF

Table 5.1.13 Chemistry - Glucose (mg/dL) - SAF
Table 5.1.14 Chemistry - HDL (mg/dL) - SAF
Table 5.1.15 Chemistry - LDL (mg/dL) - SAF

, \_\_\_ (...**g**, a\_,



Study : 105


Date: 19JAN2023

Table 5.1.16 Chemistry - Phosphorus (mg/dL) - SAF Table 5.1.17 Chemistry - Potassium (mmol/L) - SAF Table 5.1.18 Chemistry - Total Bilirubin (mg/dL) - SAF Table 5.1.19 Chemistry - Sodium (mmol/L) - SAF Table 5.1.20 Chemistry - Total Protein (g/dL) - SAF Table 5.1.21 Chemistry - Triglycerides (mg/dL) - SAF Table 5.1.22 Chemistry - Uric acid (mg/dL) - SAF Table 5.1.23 Hematology - Hematocrit (%)- SAF Table 5.1.24 Hematology - Hemoglobin (g/dL) - SAF Table 5.1.25 Hematology - MCV (fL) - SAF Table 5.1.26 Hematology - MCHC (g/L) - SAF Table 5.1.27 Hematology - Platelet count (x10<sup>3</sup> μL) - SAF Table 5.1.28 Hematology - RBC (x10<sup>6</sup> μL) - SAF Table 5.1.29 Hematology - WBC (x10^3 µL) - SAF Table 5.1.30 Hematology - Basophils (x10^3 µL) - SAF Table 5.1.31 Hematology - Eosinophils (x10<sup>3</sup> μL) - SAF Table 5.1.32 Hematology - Lymphocytes (x10<sup>3</sup> μL) - SAF Table 5.1.33 Hematology - Monocytes (x10^3 µL) - SAF Table 5.1.34 Hematology - Neutrophils (x10^3 µL) - SAF Table 5.1.35 Coagulation - INR - SAF Table 5.1.36 Coagulation - Prothrombine time (s) - SAF Table 5.1.37 Coagulation - aPTT (s) - SAF




Date: 19JAN2023

Table 5.1.38 Urine analysis – Color and appearance – SAF

| | | Fed | Fasting |
|-------------------|------|--------------|--------------|
| | | (n=xx) | (n=xx) |
| Baseline (Day -1) | | | |
| Total no-missing | n | xx | xx |
| Limpid | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Cloudy | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Hematuria | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Missing | n | xx | xx |
| 24 hours | | | |
| Total no-missing | n | xx | xx |
| Limpid | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Cloudy | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Hematuria | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Missing | n | xx | xx |
| 312 hours | | | |
| Total no-missing | n | xx | xx |
| Limpid | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Cloudy | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Hematuria | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Missing | n | xx | xx |




Date: 19JAN2023

Table 5.1.39 Urine Analysis – ph - SAF

| | | Fed | Fasting |
|-------------------|----------------|-------------------|-------------------|
| | | (n=xx) | (n=xx) |
| Baseline (Day -1) | n | xx | XX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 24 hours | n | xx | XX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | xx | xx |
| 312 hours | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1,Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (Min,Max) | (xx.x, xx.x) | (xx.x, xx.x) |
| | Missing | XX | xx |

Same table format as table 5.1.39:

Table 5.1.40 Urine analysis - Specific gravity - SAF




Date: 19JAN2023

Table 5.1.41 Urine Analysis - Glucose - SAF

| | | Fed | Fasting |
|-------------------|------|--------------|--------------|
| | | (n=xx) | (n=xx) |
| Baseline (Day -1) | | | |
| Total no-missing | n | xx | xx |
| Negative | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Trace | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| 1+ | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| 2+ | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| 3+ | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Other | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Missing | n | xx | xx |
| 24 hours | | | |
| Total no-missing | n | xx | xx |
| Negative | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Trace | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| 1+ | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| 2+ | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| 3+ | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Other | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Missing | n | xx | xx |
| 312 hours | | | |
| Total no-missing | n | xx | xx |
| Negative | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Trace | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| 1+ | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| 2+ | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| 3+ | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |




Date: 19JAN2023

| | | Fed | Fasting |
|---------|------|--------------|--------------|
| | | (n=xx) | (n=xx) |
| Other | n(%) | xx.x (xx.x%) | xx.x (xx.x%) |
| Missing | n | xx | xx |

Same table format as table 5.1.41:

Table 5.1.42 Urine Analysis – Protein – SAF

Table 5.1.43 Urine Analysis –Red blood cells – SAF

Table 5.1.44 Urine Analysis – Leukocytes – SAF

Table 5.1.45 Urine Analysis – Ketones – SAF

Table 5.1.46 Urine Analysis –Bilirubin – SAF

Table 5.1.47 Urine Analysis – Urobilinogen – SAF

Table 5.1.48 Urine Analysis – Nitrite - SAF



Study : 105 Version: 1.0

Date: 19JAN2023

# 10.5.2 Physical examination - SAF

| Table 5.2 | 2.1 Physical ex | kamination - S | AF | |
|---|---|---|---|---|
| | F | ed | Fas | ting |
| | (n: | =xx) | (n= | exx) |
| | Total no- | Name | Total no- | Nama |
| | missing<br>n | Normal<br>n (%) | missing<br>n | Normal<br>n (%) |
| Overall appropriate | " | 11 (70) | | 11 (70) |
| Overall appearance | | | | |
| Baseline (day -1) | XX | xx (xx.x%) | XX | xx (xx.x%) |
| 24 hours | xx | xx (xx.x%) | xx | xx (xx.x%) |
| 312 hours | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Skin | | | | |
| Day1 | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Head | | | | |
| Eyes and Throat | | | | |
| Thyroid | | | | |
| Lungs | | | | |
| Cardiovascular system | | | | |
| Abdomen (Liver/spleen) | | | | |
| Extremities | | | | |



Study: 105


Date: 19JAN2023

| Fe | ed | Fas | Fasting |
|-----------|--------|-----------|---------|
| (n= | =xx) | (n=xx) | |
| Total no- | | Total no- | |
| missing | Normal | missing | Normal |
| n | n (%) | n | n (%) |

Neurological

• • •



Study : 105


Date: 19JAN2023

## 10.5.3 C-SSRS

Table 5.3.1 C-SSRS - SAF

| | | Fed | Fasting |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| C-SSRS (Screening (day -28 to -2) and Baseline (day -1)) | | . , | · , , |
| Total no-missing | n | xx | XX |
| Suicidal Ideation or Behavior | n (%) | xx (xx.x%) | xx (xx.x%) |
| Suicidal Ideation | n (%) | xx (xx.x%) | xx (xx.x%) |
| Wish to dead | n (%) | xx (xx.x%) | xx (xx.x%) |
| Non-specific active suicidal thoughts | n (%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with any methods (not plan) without intent to | n (%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with some intent to act, without specific plan | n (%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with specific plan and intent | n (%) | xx (xx.x%) | xx (xx.x%) |
| Suicidal Behavior | n (%) | xx (xx.x%) | xx (xx.x%) |
| Preparatory acts or behavior | n (%) | xx (xx.x%) | xx (xx.x%) |
| Aborted attempt | n (%) | xx (xx.x%) | xx (xx.x%) |
| Interrupted attempt | n (%) | xx (xx.x%) | xx (xx.x%) |
| Non-fatal suicide attempt | n (%) | xx (xx.x%) | xx (xx.x%) |
| Self-injorious behavior without suicidal intent | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| C-SSRS (24 hours) | | | |
| Total no-missing | n | xx | xx |
| Suicidal Ideation or Behavior | n (%) | xx (xx.x%) | xx (xx.x%) |
| Suicidal Ideation | n (%) | xx (xx.x%) | xx (xx.x%) |
| Wish to dead | n (%) | xx (xx.x%) | xx (xx.x%) |
| Non-specific active suicidal thoughts | n (%) | xx (xx.x%) | xx (xx.x%) |



Study : 105


Date: 19JAN2023

Fed **Fasting** (n=xx)(n=xx) Active suicidal ideation with any methods (not plan) without intent to n (%) xx (xx.x%) xx (xx.x%) act Active suicidal ideation with some intent to act, without specific plan n (%) xx (xx.x%) xx (xx.x%) Active suicidal ideation with specific plan and intent n (%) xx (xx.x%) xx (xx.x%) Suicidal Behavior n (%) xx (xx.x%) xx (xx.x%) Preparatory acts or behavior n (%) xx (xx.x%) xx (xx.x%) Aborted attempt n (%) xx (xx.x%) xx (xx.x%) Interrupted attempt n (%) xx (xx.x%) xx (xx.x%) Non-fatal suicide attempt n (%) xx (xx.x%) xx (xx.x%) Completed suicide n (%) xx (xx.x%) xx (xx.x%) Self-injorious behavior without suicidal intent xx (xx.x%) xx (xx.x%) n (%) Missing XX XX n C-SSRS (312 hours) Total no-missing XX n XX Suicidal Ideation or Behavior n (%) xx (xx.x%) xx (xx.x%) Suicidal Ideation n (%) xx (xx.x%) xx (xx.x%) Wish to dead n (%) xx (xx.x%) xx (xx.x%) Non-specific active suicidal thoughts n (%) xx (xx.x%) xx (xx.x%) Active suicidal ideation with any methods (not plan) without intent to n (%) xx (xx.x%) xx (xx.x%) act Active suicidal ideation with some intent to act, without specific plan n (%) xx (xx.x%) xx (xx.x%) Active suicidal ideation with specific plan and intent n (%) xx (xx.x%) xx (xx.x%) Suicidal Behavior n (%) xx (xx.x%) xx (xx.x%) Preparatory acts or behavior n (%) xx (xx.x%) xx (xx.x%) Aborted attempt n (%) xx (xx.x%) xx (xx.x%) Interrupted attempt n (%) xx (xx.x%) xx (xx.x%)



Study : 105


Date: 19JAN2023

| | | Fed<br>(n=xx) | Fasting<br>(n=xx) |
|---|---|---|---|
| Non-fatal suicide attempt | n (%) | xx (xx.x%) | xx (xx.x%) |
| Completed suicide | n (%) | xx (xx.x%) | xx (xx.x%) |
| Self-injorious behavior without suicidal intent | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx |
| C-SSRS (24 hours and 312 hours) | | | |
| Total no-missing | n | xx | xx |
| Suicidal Ideation or Behavior | n (%) | xx (xx.x%) | xx (xx.x%) |
| Suicidal Ideation | n (%) | xx (xx.x%) | xx (xx.x%) |
| Wish to dead | n (%) | xx (xx.x%) | xx (xx.x%) |
| Non-specific active suicidal thoughts | n (%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with any methods (not plan) without intent to act | n (%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with some intent to act, without specific plan | n (%) | xx (xx.x%) | xx (xx.x%) |
| Active suicidal ideation with specific plan and intent | n (%) | xx (xx.x%) | xx (xx.x%) |
| Suicidal Behavior | n (%) | xx (xx.x%) | xx (xx.x%) |
| Preparatory acts or behavior | n (%) | xx (xx.x%) | xx (xx.x%) |
| Aborted attempt | n (%) | xx (xx.x%) | xx (xx.x%) |
| Interrupted attempt | n (%) | xx (xx.x%) | xx (xx.x%) |
| Non-fatal suicide attempt | n (%) | xx (xx.x%) | xx (xx.x%) |
| Completed suicide | n (%) | xx (xx.x%) | xx (xx.x%) |
| Self-injorious behavior without suicidal intent | n (%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | XX | XX |



Study: 105
Date: 19JAN2023

## 10.6 Concomitant medication

Table 6.1.1 Previous concomitant medication

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Previous concomitant medication | | | | |
| Total no missing | n | xx | XX | XX |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | xx |
| ACT classification name | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

The concomitant medication will be presented by using the WHOdrug dictionary version 2021.

Table 6.1.2 Concomitant medication during study

| | | Total subjects | Fed | Fasting |
|---|---|---|---|---|
| | | (n=xx) | (n=xx) | (n=xx) |
| Concomitant medication during study | | | | |
| Total no missing | n | xx | xx | xx |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Indication:* | | | | |
| AE | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Medical History | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | n | xx | xx | XX |
| ACT classification name | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

The concomitant medication will be presented by using the WHOdrug dictionary version 2021.

<sup>\*</sup>More than one option per patient could be possible.



| Study: 105 |
|------------------|
| Date : 19JAN2023 |

# 10.7 Listings

## Listing 7.1.1 Discontinued subjects

| Subject ID | Fed/Fasting | Date of premature withdrawal | Reason for premature withdrawal |
|---|---|---|---|
| XX | xx | XX | XX |

## Listing 7.1.2 Protocol deviations

| Subject ID | Fed/Fasting | Description | Type of deviation | Major/Minor |
|------------|-------------|-------------|-------------------|-------------|
| xx | xx | xx | XX | xx |

## Listing 7.1.3 Subjects excluded from population analysis

| Subject ID | Fed/Fasting | SAF | PK | Reason for exclusion |
|------------|-------------|-----|----|----------------------|
| XX | XX | XX | xx | XX |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 



Study : 105


Date : 19JAN2023

## Listing 7.1.4 Baseline data

| Subject ID | Fed/Fasting | Age (years) | Sex | BMI (Kg/m²) |
|------------|-------------|-------------|-----|-------------|
| xx | xx | xx | xx | xx |

## Listing 7.1.5 Prior concomitant medication

| Subject ID | Fed/Fasting | ACT level 4 <sup>1</sup> | Dose | Unit | Route | Date start | Date end | Ongoing | Indication |
|---|---|---|---|---|---|---|---|---|---|
| xx | XX | xx | xx | xx | xx | xx | xx | xx | xx |

<sup>1</sup>WHOdrug dictionary version 2021.

## Listing 7.1.6 Concomitant medication during study

| Subject ID | Fed/Fasting | ACT level 4 <sup>1</sup> | Dose | Unit | Route | Date start | Date end | Ongoing | Indication |
|---|---|---|---|---|---|---|---|---|---|
| xx | XX | xx | xx | xx | xx | xx | xx | xx | xx |

<sup>1</sup>WHOdrug dictionary version 2021.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 



Study : 105


Date : 19JAN2023

## Listing 7.1.7 Adverse Events

Alternativ

e or

confound

| Subject | TEAE | Fed/Fasti | | Preferred | | | ing Corrective | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | (yes/no) | ng | System Organ Class <sup>1</sup> | Term <sup>1</sup> | Serious | Severity | Causality | causality | Action | treatment | Outcome | Date start | Date end | Ongoing |
| XX | xx | xx | xx | xx | xx | xx | xx | xx | xx | XX | xx | XX | xx | XX |

<sup>1</sup>MedDRA dictionary version 25.0.

## Listing 7.1.8 Serious adverse events

| | | | | | | Hospitalization | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | or | | Other | | |
| | | | | | | prolongation | Congenital | medically | | Significant |
| | TEAE | | | Preferred | | of existing | anomaly or | important | Life | disability / |
| Subject ID | (yes/no) | Fed/Fasting | System Organ Class <sup>1</sup> | Term <sup>1</sup> | Death | hospitalization | birth defect | event | threatening | incapacity |
| xx | xx | xx | xx | xx | XX | xx | XX | XX | xx | xx |

<sup>1</sup>MedDRA dictionary version 25.0.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 



Study: 105


Date: 19JAN2023

## Listing 7.1.9 Abnormal findings on physical examination

| Subject ID | Fed/Fasting | Visit | System | Abnormal finding |
|------------|-------------|-------|--------|------------------|
| xx | xx | xx | xx | xx |

## Listing 7.1.10 Abnormal findings on vital signs, ECG and laboratory results

| Subject ID | Fed/Fasting | Visit | Parameter | Value <sup>1</sup> | Unit <sup>1</sup> | Results <sup>2</sup> | AE | NCS/CS |
|---|---|---|---|---|---|---|---|---|
| xx | xx | xx | xx | xx | xx | xx | xx | xx |

<sup>&</sup>lt;sup>1</sup>Chemistry, Hematology, Coagulation, Vital signs and ECG parameters.

<sup>2</sup>Urine analysis parameters

## Listing 7.1.11 COVID-19 tests

| Subject ID | Fed/Fasting | Visit | Date | Result |
|------------|-------------|-------|------|--------|
| xx | xx | XX | xx | XX |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

BioClever SOPs ST 1008-07 -CONFIDENCIAL- 